CLINICAL TRIAL: NCT06690697
Title: A Single Center, Prospective, Randomized Controlled, Second-Line Clinical Study on the Combination of Toripalimab and JS004 in the Treatment for Recurrent and Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Combination of Toripalimab and JS004 Therapy for ccRCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, MD, Professor of Urology, Fudan University Cancer Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2411091-1
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: ccRCC; toripalimab; JS004; TLSs; ORR; prognosis
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — toripalimab; Axitinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TLS-negative patients with standard second-line treatment (sorafenib or axitinib) (Active Comparator): Recurrent or metastatic clear cell renal cell carcinoma patients confirmed to be TLS-negative by HE/IHC assay will be treated with standard second-line treatment (sorafenib or axitinib).
  Interventions: Drug: Axitinib; Drug: Sorafenib
- TLS-positive patients treated with standard second-line treatment (sorafenib or axitinib) (Active Comparator): Recurrent or metastatic clear cell renal cell carcinoma patients confirmed to be TLS- positive by HE/IHC assay will be treated with standard second-line treatment (sorafenib or axitinib).
  Interventions: Drug: Axitinib; Drug: Sorafenib
- TLS-negative patients treated with toripalimab and JS004 (Experimental): Recurrent or metastatic clear cell renal cell carcinoma patients confirmed to be TLS-negative by HE/IHC assay will be treated with toripalimab and JS004.
  Interventions: Drug: JS004; Drug: Toripalimab
- TLS-positive patients treated with toripalimab and JS004 (Experimental): Recurrent or metastatic clear cell renal cell carcinoma patients confirmed to be TLS- positive by HE/IHC assay will be treated with toripalimab and JS004.
  Interventions: Drug: JS004; Drug: Toripalimab

INTERVENTIONS:
Drug: JS004 — 200 mg, ivdrip, D1, Q3W, each 21 days as a treatment cycle
  Arms: TLS-negative patients treated with toripalimab and JS004; TLS-positive patients treated with toripalimab and JS004
Drug: Toripalimab — 240 mg, ivdrip, D1, Q3W, each 21 days as a treatment cycle
  Arms: TLS-negative patients treated with toripalimab and JS004; TLS-positive patients treated with toripalimab and JS004
Drug: Axitinib — 5 mg, po, bid, each 21 days as a treatment cycle
  Arms: TLS-negative patients with standard second-line treatment (sorafenib or axitinib); TLS-positive patients treated with standard second-line treatment (sorafenib or axitinib)
Drug: Sorafenib — 0.4 g, po, bid, each 21 days as a treatment cycle
  Arms: TLS-negative patients with standard second-line treatment (sorafenib or axitinib); TLS-positive patients treated with standard second-line treatment (sorafenib or axitinib)

SUMMARY:
This study is a single center, prospective, randomized controlled phase II clinical trial aimed at examining the efficacy and safety of the combination of toripalimab and JS004 versus standard therapy for second-line treatment of recurrent and metastatic clear cell renal cell carcinoma patients. The study population consists of recurrent and metastatic renal cell carcinoma patients who have undergone radical operation and have been histologically confirmed as clear cell subtype. The subjects will receive JS004 combined with toripalimab or standard second-line treatment. The main endpoint of this study is the Overall Response Rate (ORR). In addition, we will explore the ORR, Disease Control Rate (DCR), Progression-Free Survival (PFS), and Overall Survival (OS) of different subgroups of tertiary lymphoid structures (TLSs) presence, location, density, quantity, and maturity in primary tumors. This study is a randomized controlled trial, with a total of 80 participants planned to be included, with regular follow-up for monitoring disease progression and treatment safety. The study will be conducted at Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participated in this study, signed an informed consent form, and showed good compliance;
2. Age ≥ 18 years old;
3. Local recurrence or metastatic renal cell carcinoma that has undergone curative surgical resection and has been histologically confirmed;
4. Previous treatment history of the subject: patients who have received one type of systemic therapy in the past and have progressed or become intolerant, as well as patients who have progressed within 6 months after previous adjuvant or neoadjuvant therapy;
5. Patients are required to provide postoperative tissue wax blocks for research and testing purposes, which should include both renal cancer tissue and normal kidney tissue adjacent to the cancer. Alternatively, at least 20 slices of previous surgical specimens should be provided for HE/IHC/spatial omics testing; The criteria for detecting TLS positivity are: detecting at least one CD3+/CD20+lymphocyte aggregate containing>700 cells in the tumor;
6. Have at least one measurable lesion (RECIST 1.1);
7. ECOG score 0-1;
8. The main organ functions well, and the laboratory examination indicators meet the following criteria:

(1) Blood routine examination:

* Hemoglobin (HB) ≥ 80g/L;

  ② Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Total white blood cell count ≥ 3.5 × 109/L;

  ③ Platelet count (PLT) ≥ 80 × 109/L; (2) Blood biochemistry test:
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for liver/bone metastases; ≤ 5 ULN for tumor bone metastases);

  * Serum total bilirubin (TBIL) ≤ 1.5 × ULN; ③ Serum creatinine Cr ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min; (3) Coagulation function test: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN; (4) Thyroid function: Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group) 9. Women of childbearing age must confirm their non pregnancy status before enrollment, and all enrolled subjects (male or female) should take adequate contraceptive measures throughout the entire treatment period and within 4 weeks after the end of treatment; 10. The patient voluntarily joined this study, signed an informed consent form, had good compliance, and was able to accept follow-up from the trial personnel.

Exclusion Criteria:

Patients with any of the following conditions are not eligible for inclusion in this study:

1. Known to have allergic reactions to the therapeutic drugs and/or any excipients used in this study;
2. Four weeks before the first study medication, receive systemic treatment with other anti-tumor drugs (if it has a half-life of five, it can be included in the group), or receive local anti-tumor treatment, or receive clinical investigational drug or device treatment;
3. Patients who have previously received treatment with anti BTLA or anti HVEM antibodies;
4. Subjects with standard second-line treatment and/or contraindications to the use of trastuzumab or JS004;
5. Subjects with previous or concurrent malignant tumors (excluding cured cervical cancer, basal or squamous skin cancer);
6. Active autoimmune diseases that require systemic treatment within the past 3 months, or clinically severe autoimmune disease records, or syndromes that require systemic steroids or immunosuppressants;
7. Known history of human immunodeficiency virus infection (HIV1/2 antibody positive);
8. Female participants who are pregnant, breastfeeding, or planning to become pregnant during the study period;
9. Patients with bleeding tendencies (such as active gastrointestinal ulcers) or treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues;
10. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, symptomatic interstitial lung disease, or any evidence of active pneumonia detected on chest CT scan within 4 weeks prior to the first study drug treatment;
11. According to the researcher's judgment, there are accompanying diseases that pose a serious threat to patient safety or affect the completion of the study.
12. There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the study results, as well as patients who the researcher deems unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  The number and proportion of subjects with BOR of CR or PR were calculated, and the Clopper-Pearson method was used to estimate and provide the corresponding 95 % confidence interval.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 years
  The number and proportion of subjects with BOR of CR, PR or SD were calculated, and the Clopper-Pearson method was used to estimate and provide the corresponding 95 % confidence interval.
Progression Free Survival (PFS) | 2 years
  The PFS rate and its 95 % CI were estimated by Kaplan-Meier method, the median PFS and its 95 % CI were calculated, and the Kaplan-Meier survival curve was drawn.
Overall Survival (OS) | 2 years
  The Kaplan-Meier method was used to estimate the OS rate and its 95 % CI. The median OS and its 95 % CI were calculated, and the Kaplan-Meier survival curve was drawn.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China